CLINICAL TRIAL: NCT03129438
Title: Impact on Clinical Outcome of Continuous Video-electroencephalography (cEEG) Monitoring in Patients With Disorders of Consciousness: A Randomized Controlled Trial
Brief Title: Continuous EEG Randomized Trial in Adults
Acronym: CERTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrea Rossetti, MD (Other)
Responsible Party: Sponsor-Investigator, Andrea Rossetti, MD, Associate professor, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2017_00268
Record Dates: First submitted 2017-04-17; First posted 2017-04-26 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: EEG With Periodic Abnormalities; EEG With Abnormally Slow Frequencies; Coma; Outcome, Fatal
Keywords: continuous EEG; routine EEG; prognosis
MeSH Terms: conditions — Coma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blind assessment of secondary outcomes at 6 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- continuous EEG (cEEG) (Experimental): Patients randomized to continuous EEG will be recorded with at least 21 electrodes placed according to the international 10-20 system; occasionally, a reduced montage will be allowed in patients with extensive neurosurgical scars, according to good common practice. Recordings will last a minimum of 30 and a maximum of 48 hours. During this time, one interruption to a maximum of two hours for diagnostic purposes will be allowed. Reactivity testing using auditory and nociceptive stimuli will be performed at least twice during the recording time. Recordings will be visually interpreted by certified electroencephalographers (i.e., interpretation of the automated algorithm only won't be allowed) using the 2013 American Clinical neurophysiology nomenclature; interpretations will be communicated within two hours of their completion to the treating team.
  Interventions: Diagnostic Test: continuous EEG (cEEG)
- routine EEG (rEEG) (Active Comparator): Patients randomized to routine EEG will be recorded with at least 21 electrodes placed according to the international 10-20 system; occasionally, a reduced montage will be allowed in patients with extensive neurosurgical scars, according to good common practice. Recordings will last between 20 and 30 minutes; two recordings will take place over a period of 24 to 48 hours. Reactivity testing using auditory and nociceptive stimuli will be performed once per recording. Recordings will be visually interpreted by certified electroencephalographers using the 2013 American Clinical neurophysiology nomenclature, as for the experimental intervention, and the interpretation will be communicated within two hours of its completion to the treating team.
  Interventions: Diagnostic Test: routine EEG (rEEG)

INTERVENTIONS:
Diagnostic Test: continuous EEG (cEEG) — differential use of continuous versus routine EEG
  Arms: continuous EEG (cEEG)
Diagnostic Test: routine EEG (rEEG) — differential use of continuous versus routine EEG
  Arms: routine EEG (rEEG)

SUMMARY:
Continuous video-EEG monitoring (cEEG) significantly improves seizure or status epilepticus detection in patients in intensive care units (ICUs), and is recommended for patients with consciousness impairment. cEEG is time- and resource consuming as compared to routine EEG (rEEG, lasting 20-30 minutes). While centers in North America have been using it increasingly, most European hospitals still do not have resources to comply with these guidelines. In addition, only one population-based study based on discharge diagnoses suggested that cEEG may improve patients' outcome. Current guidelines are thus based upon weak evidence and expert opinions.

Aim of the study is to assess if cEEG in adults with consciousness impairment is related to an improvement of functional outcome, and to address the prognostic role of quantitative network EEG analyses.

In this multicenter randomized controlled trial, adults with GCS inferior or equal to 11 or FOUR score inferior or equal to 12 will be randomized 1:1 to cEEG for 30-48 hours or two rEEG within 48 hours. The primary outcome will be mortality at 6 months. Secondary outcomes will blindly assess functional outcome, seizure/status epilepticus detection rate, duration of ICU stay, change in patient management (antiepileptic drug introduced, increased, or stopped, brain imaging), and reimbursement. Additionally, quantitative EEG will be assessed towards the primary outcome. 350 patients are planned to be included.

DETAILED DESCRIPTION:
Background: Continuous video-EEG monitoring (cEEG) is a non-invasive tool to monitor the electrical brain function; it significantly improves seizure or status epilepticus detection in comatose patients in intensive care units (ICUs), which often do not show any specific clinical correlates. Recently, the European Society of Intensive Care Medicine published guidelines regarding the use of cEEG in the ICUs, recommending it for most patients with consciousness disorders. cEEG is time- and resource consuming as compared to routine spot EEG (rEEG, typically lasting 20-30 minutes). While centers in North America have been using it increasingly, most European - and all Swiss - hospitals still do not have enough resources to comply with these guidelines. In addition, while the superiority of cEEG to detect non-convulsive seizures or status epilepticus is proven, only one population-based study based on discharge diagnoses suggested that cEEG may improve patients' outcome. Current guidelines are thus based upon weak evidence and expert opinions. If cEEG leads to improved patients' care remains elusive. Moreover, little attention has been drawn towards quantitative EEG information beyond visual analysis, and the impact of such information on diagnosis, treatment, and outcome remains unclear.

Aim: To assess whether the use of cEEG in patients with consciousness impairment is related to an improvement of functional outcome, and to address the prognostic role of quantitative network EEG analyses in this cohort. Also, a cost analysis will be performed.

Methods: In this multicenter randomized controlled trial, adults with a Glasgow Coma Score (GCS) inferior or equal to 11 or a FOUR score inferior or equal to 12, regardless of etiologies, will be randomized 1:1 to cEEG for 30-48 hours or two rEEG within 48 hours, interpreted in a standardized way. Patients with detected seizures in the last 36h or status epilepticus in the last 96h will be excluded, as cEEG may represent the standard of care. Demographics, etiology, Charlson Comorbidity Index, GCS, diagnosis leading to EEG, mechanical ventilation, and subsequent use of rEEG/cEEG will be collected. The primary outcome will be mortality at 6 months. Secondary outcomes will blindly assess functional outcome at 4 weeks and 6 months, as well as seizure/status epilepticus detection rate and time to detection, infections rate, duration of ICU stay, change in patient management (antiepileptic drug introduced, increased, or stopped, brain imaging), and reimbursement. Analyses will compare the two interventional groups (intention to diagnose) regarding outcome, as a whole and stratified according to etiological subgroups, and other variables of interest. Additionally, lope cross correlation and horizontal visibility graphs will be applied to compute a weighted adjacency matrix consisting of all the pairwise interdependences between EEG signals, in order to characterize the integrative and segregative characteristics of the underlying functional brain networks and compare their relationship with the primary outcome. According to a previous estimate, patients with consciousness disorders undergoing cEEG have a 75% survival rate; while patients w/o cEEG 61%. Using a power of 0.8, an α error of 0.05, and a 2-side approach, 2x174 patients would be needed to detect this significant difference in survival.

Expected impact: This study will clarify if cEEG monitoring has a significant impact on functional outcome and define its cost effectiveness, and if network EEG analysis has a role in outcome prognostication. The results of this study will have a considerable potential to influence clinical practice regarding EEG and treatment of patients with altered levels of consciousness. If results will indicate that cEEG contributes to improve outcome, this will lead to the urgent need for implementation of cEEG with consecutive substantial impact on health care and resource allocation in larger Swiss and European hospitals.

ELIGIBILITY:
Inclusion Criteria:

* In-patients aged ≥18 years, treated in an ICU or intermediate care unit
* Alteration of mental state of any etiology (i.e., primarily cerebral or not), with Glasgow-coma scale inferior or equal to 11 or FOUR score inferior or equal to 12.
* Need of an EEG to exclude seizures or SE, or to evaluate prognosis as per the treating physician or the consulting neurologist.
* Informed consent obtained for research in emergency situation according to Human Research Act (HRA) art 30-31 at the time of inclusion

Exclusion Criteria:

* Clinical and/or electrographic status epilepticus < 96h before randomization
* Clinical and/or electrographic seizure < 36h before randomization
* Palliative care situation, in which detection of SE or seizures would not have any impact on the patient's care.
* High likelihood of needing a surgical intervention or an invasive diagnostic procedure within the next 48 hours according to the treating physician (as this would require cEEG removal).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

PRIMARY OUTCOMES:
Mortality | 6 months
  Fatality rate

SECONDARY OUTCOMES:
Functional outcome 1 | 4 weeks, 6 months
  Functional outcome using the modified Rankin Scale (mRS) (ordinal)
Functional outcome 2 | 4 weeks, 6 months
  Functional outcome using the Cerebral Performance Categories (CPC) (ordinal)
Work/School | 4 weeks, 6 months
  Assessment of ability to go back to work/school if previously working/at school (proportion)
Seizure detection rate | within 60 hours
  Seizure detection rate (proportion)
Status Epilepticus detection rate | within 60 hours
  Status Epilepticus detection rate (proportion)
Time to detection of seizure | within 60 hours
  Time to detection of seizure after the start of EEG recording (continuous variable)
Time to detection of status epilepticus | within 60 hours
  Time to detection of status epilepticus after the start of EEG recording (continuous variable)
Presence of clinical signs of seizures | within 60 hours
  Presence of clinical signs of seizures (continuous variable)
Detection of interictal epileptiform features | within 60 hours
  Detection of interictal epileptiform features (categorical)
Rate of Infections | 4 weeks
  Rate of in-hospital infections requiring antibiotic treatment at 4 weeks after first EEG (proportion)
Need of mechanical ventilation | 4 weeks
  Need of mechanical ventilation after first EEG (proportion variable)
Duration of mechanical ventilation | 4 weeks
  Duration of mechanical ventilation after first EEG (continuous variable)
Duration of ICU and hospital stay | 4 weeks, 6 months
  Duration of ICU and hospital stay (continuous variable)
Patient destination | 4 weeks, 6 months
  Patient destination after acute facility (home, rehab, nursing home, other; categorical)
Change in clinical patients' management | 60 hours
  Change in clinical patient management (i.e., antiepileptic drugs (AED) introduced or stopped, AED increased or decreased, brain imaging procedure order) occurring during the 60 hours following the start of the first EEG (categorical).
Correlation between quantitative EEG and primary outcome | 6 months
  Correlation between quantitative EEG and primary outcome
Hospitalization costs | 6 months
  Global hospitalization costs intended as amount billed for each patient's acute hospital stay, assessed through the billing department of each hospital (continuous variable - stratified by site)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea O Rossetti, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (4):
- Switzerland (4):
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud
  - Hôpital du Valais - Site Hôpital de Sion, Sion, Valais
  - Universitätsspital, Basel
  - Inselspital, Bern

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Urbano V, Alvarez V, Schindler K, Ruegg S, Ben-Hamouda N, Novy J, Rossetti AO. Continuous versus routine EEG in patients after cardiac arrest: Analysis of a randomized controlled trial (CERTA). Resuscitation. 2022 Jul;176:68-73. doi: 10.1016/j.resuscitation.2022.05.017. Epub 2022 May 30. PMID 35654226
- [Derived] Urbano V, Novy J, Alvarez V, Schindler K, Ruegg S, Rossetti AO. EEG recording latency in critically ill patients: Impact on outcome. An analysis of a randomized controlled trial (CERTA). Clin Neurophysiol. 2022 Jul;139:23-27. doi: 10.1016/j.clinph.2022.04.003. Epub 2022 Apr 18. PMID 35490437
- [Derived] Urbano V, Novy J, Schindler K, Ruegg S, Alvarez V, Zubler F, Oddo M, Lee JW, Rossetti AO. Continuous versus routine EEG in critically ill adults: reimbursement analysis of a randomised trial. Swiss Med Wkly. 2021 Mar 16;151:w20477. doi: 10.4414/smw.2021.20477. eCollection 2021 Mar 15. PMID 33793960
- [Derived] Guinchard M, Warpelin-Decrausaz L, Schindler K, Ruegg S, Oddo M, Novy J, Alvarez V, Rossetti AO. Informed consent in critically ill adults participating to a randomized trial. Brain Behav. 2021 Feb;11(2):e01965. doi: 10.1002/brb3.1965. Epub 2020 Dec 3. PMID 33271000
- [Derived] Rossetti AO, Schindler K, Sutter R, Ruegg S, Zubler F, Novy J, Oddo M, Warpelin-Decrausaz L, Alvarez V. Continuous vs Routine Electroencephalogram in Critically Ill Adults With Altered Consciousness and No Recent Seizure: A Multicenter Randomized Clinical Trial. JAMA Neurol. 2020 Oct 1;77(10):1225-1232. doi: 10.1001/jamaneurol.2020.2264. PMID 32716479